CLINICAL TRIAL: NCT01087983
Title: A Phase 1 Trial of Lapatinib in Combination With 1) Sirolimus or 2) Metformin in Advanced Cancer
Brief Title: Lapatinib With Sirolimus or Metformin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0743; NCI-2011-00563 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-03-15; First posted 2010-03-16 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-11

CONDITIONS: Advanced Cancers
Keywords: Metastatic cancer; Lapatinib; Tykerb; Metformin; Glucophage; Sirolimus; Rapamune
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Lapatinib; Sirolimus; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lapatinib + Sirolimus (Experimental): Lapatinib starting oral dose of 500 mg daily for 21 day cycle. Sirolimus starting oral dose 1 mg daily.
  Interventions: Drug: Lapatinib; Drug: Sirolimus
- Lapatinib + Metformin (Experimental): Lapatinib starting oral dose of 500 mg daily for 21 day cycle. Metformin Starting oral dose 1000 mg daily.
  Interventions: Drug: Lapatinib; Drug: Metformin

INTERVENTIONS:
Drug: Lapatinib — Starting oral dose of 500 mg daily for 21 day cycle.
  Other Names: Tykerb; GW572016
Drug: Sirolimus — Starting oral dose 1 mg daily.
  Other Names: Rapamune
  Arms: Lapatinib + Sirolimus
Drug: Metformin — Starting oral dose 1000 mg daily.
  Other Names: Glucophage
  Arms: Lapatinib + Metformin

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of 2 different combinations of drugs that can be given to patients with advanced cancer. The first combination of drugs is Tykerb (lapatinib) and Rapamune (sirolimus), and the second combination is lapatinib and Glucophage (metformin). The safety of these drug combinations will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Lapatinib is designed to prevent or slow down the growth of cancer cells by blocking 2 proteins on the surface of the cancer cell, which are HER 1 and HER 2 receptors.

Sirolimus is designed to block a protein called mammalian target of rapamycin (mTOR) (a protein that is thought to cause cancer cells to grow) inside the cancer cell. This may interfere with the growth or spread of cancer cells or possibly kill the cancer cells.

Metformin was designed to treat patients with diabetes. It may be able to block mTOR and slow the growth of tumors.

Study Drug Groups:

If you are found to be eligible to take part in this study, your doctor will decide if you will receive lapatinib with metformin or lapatinib with sirolimus. Once it is decided which combination you will receive, you will be assigned to a dose level based on when you join the study.

Up to 7 dose levels of lapatinib with sirolimus will be tested. Up to 6 dose levels of lapatinib with metformin will be tested. Three (3) to 6 participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of the combination of lapatinib with either sirolimus or metformin is found.

Once the highest tolerated dose of the combination of lapatinib with either sirolimus or metformin is found, 14 participants with the tumor type that has responded to the study drug combination will receive the study drugs at that dose level.

Study Drug Administration:

Each study "cycle" is 28 days.

You will take lapatinib by mouth 1 time each day. You should take it at about the same time each day on an empty stomach with a cup (about 8 ounces) of water, 1 hour before and 2 hours after a meal.

If you are also taking metformin, you will take it by mouth 1 time every day. You should take it at about the same time each day with a meal and cup of water (about 8 ounces).

If you are also taking sirolimus, you will take it by mouth 1 time every day. You should take it at about the same time each day on an empty stomach with a cup of water, 1 hour before and 2 hours after a meal.

Study Visits:

At every study visit, you will be asked about any current health conditions you have, any other drugs you are taking, and if you have experienced any side effects.

On about Days 1, 8, and 15 of Cycle 1, blood (about 2 teaspoons) will be drawn for routine tests.

On about Day 1 Cycle 1, urine will be collected for routine tests.

On about Day 1 of Cycles 2 and beyond:

* You will have a physical exam.
* Blood (about 2 teaspoons) and urine will be collected for routine tests.

Every 6 weeks, you will have a blood (about 1 teaspoon) drawn or urine collected for pregnancy test if you are able to become pregnant.

Every 8 weeks for the first 4 cycles, you will have an x-ray, CT scan, MRI scan, and/or PET/CT scan to check the status of the disease. If the study doctor thinks it is needed, they will be performed more often. After 4 cycles you will have an x-ray, CT scan, MRI scan, and/or PET/CT scan every 8 - 12 weeks as your study if the study doctor feels it is appropriate.

Length of Study:

You may stay on study for as long as you are benefitting. You will be taken off study if you experience intolerable side effects, the study doctor thinks it is in your best interest, or the disease gets worse.

This is an investigational study. Sirolimus is FDA approved and commercially available as an anti-rejection drug for kidney transplant recipients. Lapatinib is FDA approved and commercially available for the treatment of advanced breast cancer. Metformin is FDA approved and commercially available for the treatment of diabetes mellitus. The combination of these drugs to treat advanced cancer is investigational.

Up to 106 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced or metastatic cancer that is refractory to standard therapy, relapsed after standard therapy, or who have no standard therapy available that improves survival by at least three months.
2. Patients must be at least 3 weeks beyond their previous cytotoxic treatment. Patient must wait at least 5 half-lives or 3 weeks, whichever is shorter, from their previous targeted or biologic therapy; In addition, patients must be at least 3 weeks beyond the last session of radiation therapy or major surgery. Local palliative radiation therapy that is not delivered to all target lesions is allowed immediately before or during treatment.
3. Eastern Cooperative Oncology Group (ECOG) performance status should be less or equal to 3
4. Patients must have normal organ and marrow function defined as: absolute neutrophil count (ANC) >/= 750/mL; platelets >/= 50,000/mL; creatinine </= 2x upper limit of normal (ULN) for the Sirolimus Arm and creatinine < 1.5 mg/dl for the Metformin arm; total bilirubin </=2.0 (For patients with Gilbert syndrome, bilirubin level > 2 could will be allowed on study if the hyperbilirubinemia is believed to be secondary only to the Gilbert syndrome); ALT (SGPT) </= 5x ULN; Exception for patients with liver metastasis: total bilirubin </= 3x ULN; ALT (SGPT) </= 8x ULN.
5. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 30 days after the last dose
6. Patients must be able to understand and be willing to sign a written informed consent document
7. Patients with treated brain metastases are allowed in both arms of the study.

Exclusion Criteria:

1. Uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, uncontrolled asthma, need for hemodialysis, need for ventilatory support.
2. Pregnant or lactating women.
3. History of hypersensitivity to Lapatinib or any component of the formulation.
4. Patients who have malabsorption syndrome
5. Patients with class III or IV congestive heart failure as defined by New York Heart Association functional classification system
6. Patients unwilling or unable to sign informed consent document
7. History of hypersensitivity to Sirolimus or any component of the formulation (for Lapatinib and Sirolimus arm only)
8. History of hypersensitivity to metformin or any component of the formulation (for Lapatinib and Metformin arm only)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2010-03; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Lapatinib in Combination with Sirolimus or Metformin | 21 day cycle
  MTD is defined as the highest dose studied in which the incidence of dose-limiting toxicity (DLT) is less than 33%.

CONTACTS AND LOCATIONS:
Overall Officials: Filip Janku, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org